CLINICAL TRIAL: NCT03504943
Title: Timing of Intradialytic Exercise and Its Impact on Intradialytic Hypotension: a Randomized Crossover Study
Brief Title: Timing of Intradialytic Exercise and Its Impact on Intradialytic Hypotension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: University of Alberta (Other); University of Calgary (Other)
Responsible Party: Principal Investigator, Clara Bohm, Associate Professor, Nephrologist, University of Manitoba
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: HS21703 (B2018:035)
Record Dates: First submitted 2018-04-12; First posted 2018-04-20 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Intradialytic Hypotension; Hemodialysis-Induced Symptoms
Keywords: Exercise; Hemodialysis; Intradialytic hypotension
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Intradialytic Exercise (Active Comparator): Intradialytic cycling will occur in the first half of hemodialysis treatment
  Interventions: Other: Early Intradialytic Exercise
- Late Intradialytic Exercise (Experimental): Intradialytic cycling will occur in the second half of hemodialysis treatment
  Interventions: Other: Late Intradialytic Exercise

INTERVENTIONS:
Other: Early Intradialytic Exercise — Timing of intradialytic exercise first half of HD
  Arms: Early Intradialytic Exercise
Other: Late Intradialytic Exercise — Timing of intradialytic exercise second half of HD
  Arms: Late Intradialytic Exercise

SUMMARY:
The objective of this study is to compare the rate of low blood pressure events (Intradialytic Hypotension: IDH) when intradialytic exercise is performed in the first half of the hemodialysis (HD) session as compared to that when intradialytic exercise is performed in the second half of the HD session. The investigators expect that there will be little to no difference in occurrence of IDH episodes between the two time periods based on the experience of the 3 centres and imaging studies of the heart with exercise in HD.

DETAILED DESCRIPTION:
Intradialytic hypotension (IDH) is a common complication during hemodialysis, occurring in 20-30% of HD treatments. IDH can cause unpleasant symptoms and lead to decline in residual kidney function, vascular access thrombosis, ischemic damage to white matter of the brain, volume overload, increased risk of cardiovascular events and increased mortality risk.

Intradialytic exercise has been shown to improve physical function, health-related quality of life and cardiac function. Initial concerns regarding the potential for intradialytic exercise to increase the rate of IDH have been mitigated by multiple interventional studies in which intradialytic exercise has been shown to be safe with minimal adverse effects. However, concerns regarding the potential of intradialytic exercise to increase frequency of IDH if exercise is performed in second half of HD remain.

No study has specifically compared the frequency IDH episodes when exercise is performed during second half of HD as compared to that when exercise is performed during the first half of a HD session to fully characterize the effect of timing of intradialytic exercise and its effect on IDH.

The investigators aim to address this knowledge gap with a crossover study examining the rate of IDH when individuals in a clinical intradialytic cycling program exercise during the first half of their hemodialysis session as compared with the IDH rate when exercise is performed during the second half of hemodialysis.

To facilitate study implementation and optimize use of exercise resources and equipment, participants at each site will be randomly split into 2 groups. Group 1 will perform 2 weeks of their usual intradialytic cycling (6 sessions) during the first half of their usual HD and then perform 2 weeks of intradialytic cycling (6 sessions) during the second half of their usual HD. Group 2 will perform the intervention in reverse order to Group 1. No washout period is required as there is no biological plausibility for carry over effect. However, as participation in the cycling program is voluntary, some participants choose not to exercise during some of their HD sessions. The investigators will monitor these non-cycling sessions for IDH as well and will compare IDH rate in these non-exercise sessions with IDH rate during sessions when intradialytic exercise was performed, if numbers allow.

Participants will perform their usual duration and intensity of intradialytic cycling at each HD session as per standard clinical intradialytic cycling protocol procedures in each unit. Prescribed exercise time and intensity will remain unchanged over the course of the study.

The investigators will attempt to keep dialysate composition, dialyzer, dialysate temperature, HD access, dialysis duration and medications unchanged over the course of the study, but will not intervene/interfere with usual clinical care. The research assistant will record any changes to dialysis prescription related to routine clinical care on a weekly basis.

Baseline demographic and clinical data will be collected from the hemodialysis chart. This will include age, sex, race, time on hemodialysis, hemodialysis access, dialysis vintage, comorbidities (including hypertension, diabetes, congestive heart failure and ischemic heart disease), amount of fluid removed at each HD, hemoglobin, Kt/V (dialysis efficacy), medications and blood work results as measured on last monthly bloodwork.

The investigators will use the initial BP measurement obtained once the patient has commenced HD (i.e. patient "hooked up" and blood present in both venous and arterial lines) for the baseline BP. Blood pressure (BP) will be measured as per routine procedures used in the participants' HD units (usual arm/leg, usual BP cuff). Pre and post HD BP will be collected as per usual HD Unit practice. During HD, BP will be collected more frequently than the usual routine (q30 min) at q15min intervals or more frequently when clinically indicated based on patient symptoms or status. This timing will be pre-programmed into HD machines to minimize work for bedside HD nurses. However, bedside HD nurses will need to record each measurement on the HD run sheet.

ELIGIBILITY:
Inclusion Criteria:

* adult (>= 18 years old), receiving three times per week chronic in-centre hemodialysis, current active participant in clinical intradialytic cycling program offered at each study site, able to communicate in English, able to provide written consent

Exclusion Criteria:

* dialysis frequency not three times per week

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2018-07-09 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Difference in the rate of IDH (episodes of hypotension per 100 hours of HD) between the 2 study time periods (early and late intradialytic exercise) | 4 weeks
  IDH will be defined as a composite of >= 20 mmHg drop from baseline bp or a drop in systolic BP to <90 mmHg

SECONDARY OUTCOMES:
Difference in rate of IDH (episodes of hypotension per 100 hours of HD) between the 2 study time periods AND associated symptoms OR requiring intervention by bedside nurse | 4 weeks
  IDH as defined by a >20 mmHg drop from baseline BP. IDH associated symptoms as follows: abdominal discomfort, yawning, sighing, nausea, vomiting, muscle cramps, restlessness, dizziness or fainting, and anxiety
Difference in frequency and severity of dialysis-related symptoms as measured by the Dialysis Symptom Index between exercise performed in the first and second half of HD sessions. | 4 weeks
  Frequency and severity of symptoms will be measured using the symptom burden score as measured by the Dialysis Symptom Index (DSI). The DSI is a 30-item self-administered questionnaire with low administrative burden that measures the presence (yes/no) and severity (5 point Likert-scale) of common symptoms in HD patients (cramping, nausea, dizziness, fatigue, chest pain and shortness of breath) and has been shown to be reliable and valid. Participants will complete the DSI at time of consent and then weekly at the end of the midweek HD session for the duration of the study
Difference in time for recovery post-dialysis between the 2 study time periods (early and late intradialytic exercise) | 4 weeks
  Participants will be asked to answer the question "Approximately how much time does it take to recover from a dialysis session?" at each study assessment. Answers will be recorded in minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Clara Bohm, MD, MPH, Principal Investigator — University of Manitoba; Jennifer MacRae, MD,MSc, Principal Investigator — University of Calgary; Stephanie Thompson, MD, PhD, Principal Investigator — University of Alberta
Locations (3):
- Canada (3):
  - University of Calgary Cumming School of Medicine Department of Internal Medicine, Calgary, Alberta
  - University of Alberta Department of Internal Medicine, Edmonton, Alberta
  - University of Manitoba Department of Internal Medicine, Winnipeg, Manitoba

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Damasiewicz MJ, Polkinghorne KR. Intra-dialytic hypotension and blood volume and blood temperature monitoring. Nephrology (Carlton). 2011 Jan;16(1):13-8. doi: 10.1111/j.1440-1797.2010.01362.x. PMID 21175972
- [Background] Daugirdas JT, Blake PG, Ing TS. Handbook of Dialysis. Lippincott Williams & Wilkins; 2014.
- [Background] K/DOQI Workgroup. K/DOQI clinical practice guidelines for cardiovascular disease in dialysis patients. Am J Kidney Dis. 2005 Apr;45(4 Suppl 3):S1-153. No abstract available. PMID 15806502
- [Background] Hayes W, Hothi DK. Intradialytic hypotension. Pediatr Nephrol. 2011 Jun;26(6):867-79. doi: 10.1007/s00467-010-1661-4. Epub 2010 Oct 22. PMID 20967553
- [Background] Gul A, Miskulin D, Harford A, Zager P. Intradialytic hypotension. Curr Opin Nephrol Hypertens. 2016 Nov;25(6):545-550. doi: 10.1097/MNH.0000000000000271. PMID 27606498
- [Background] Rocco MV, Burkart JM. Prevalence of missed treatments and early sign-offs in hemodialysis patients. J Am Soc Nephrol. 1993 Nov;4(5):1178-83. doi: 10.1681/ASN.V451178. PMID 8305644
- [Background] Iseki K, Miyasato F, Tokuyama K, Nishime K, Uehara H, Shiohira Y, Sunagawa H, Yoshihara K, Yoshi S, Toma S, Kowatari T, Wake T, Oura T, Fukiyama K. Low diastolic blood pressure, hypoalbuminemia, and risk of death in a cohort of chronic hemodialysis patients. Kidney Int. 1997 Apr;51(4):1212-7. doi: 10.1038/ki.1997.165. PMID 9083288
- [Background] Shoji T, Tsubakihara Y, Fujii M, Imai E. Hemodialysis-associated hypotension as an independent risk factor for two-year mortality in hemodialysis patients. Kidney Int. 2004 Sep;66(3):1212-20. doi: 10.1111/j.1523-1755.2004.00812.x. PMID 15327420
- [Background] Momeni A, Nematolahi A, Nasr M. Effect of intradialytic exercise on echocardiographic findings in hemodialysis patients. Iran J Kidney Dis. 2014 May;8(3):207-11. PMID 24878943
- [Background] Heiwe S, Jacobson SH. Exercise training for adults with chronic kidney disease. Cochrane Database Syst Rev. 2011 Oct 5;2011(10):CD003236. doi: 10.1002/14651858.CD003236.pub2. PMID 21975737
- [Background] Leung K, Quinn RR, Ravani P, et al. Exercise Training During Hemodialysis is not Associated with Intradialytic Hypotension. Canadian Society of Nephrology Annual Meeting; April 25, 2017, 2014; Vancouver, B.C.
- [Background] Giannaki CD, Stefanidis I, Karatzaferi C, Liakos N, Roka V, Ntente I, Sakkas GK. The effect of prolonged intradialytic exercise in hemodialysis efficiency indices. ASAIO J. 2011 May-Jun;57(3):213-8. doi: 10.1097/MAT.0b013e318215dc9e. PMID 21412149
- [Background] Farese S, Budmiger R, Aregger F, Bergmann I, Frey FJ, Uehlinger DE. Effect of transcutaneous electrical muscle stimulation and passive cycling movements on blood pressure and removal of urea and phosphate during hemodialysis. Am J Kidney Dis. 2008 Oct;52(4):745-52. doi: 10.1053/j.ajkd.2008.03.017. Epub 2008 May 19. PMID 18487001
- [Background] Rhee SY, Song JK, Hong SC, Choi JW, Jeon HJ, Shin DH, Ji EH, Choi EH, Lee J, Kim A, Choi SW, Oh J. Intradialytic exercise improves physical function and reduces intradialytic hypotension and depression in hemodialysis patients. Korean J Intern Med. 2019 May;34(3):588-598. doi: 10.3904/kjim.2017.020. Epub 2017 Aug 25. PMID 28838226
- [Background] Dungey M, Bishop NC, Young HM, Burton JO, Smith AC. The Impact of Exercising During Haemodialysis on Blood Pressure, Markers of Cardiac Injury and Systemic Inflammation--Preliminary Results of a Pilot Study. Kidney Blood Press Res. 2015;40(6):593-604. doi: 10.1159/000368535. Epub 2015 Nov 18. PMID 26619202
- [Background] Burton JO, Jefferies HJ, Selby NM, McIntyre CW. Hemodialysis-induced cardiac injury: determinants and associated outcomes. Clin J Am Soc Nephrol. 2009 May;4(5):914-20. doi: 10.2215/CJN.03900808. Epub 2009 Apr 8. PMID 19357245
- [Background] Burton JO, Jefferies HJ, Selby NM, McIntyre CW. Hemodialysis-induced repetitive myocardial injury results in global and segmental reduction in systolic cardiac function. Clin J Am Soc Nephrol. 2009 Dec;4(12):1925-31. doi: 10.2215/CJN.04470709. Epub 2009 Oct 1. PMID 19808220
- [Background] Flythe JE, Xue H, Lynch KE, Curhan GC, Brunelli SM. Association of mortality risk with various definitions of intradialytic hypotension. J Am Soc Nephrol. 2015 Mar;26(3):724-34. doi: 10.1681/ASN.2014020222. Epub 2014 Sep 30. PMID 25270068
- [Background] Awuah KT, Afolalu BA, Hussein UT, Raducu RR, Bekui AM, Finkelstein FO. Time to recovery after a hemodialysis session: impact of selected variables. Clin Kidney J. 2013 Dec;6(6):595-8. doi: 10.1093/ckj/sft120. Epub 2013 Sep 29. PMID 26069828
- [Background] Lindsay RM, Heidenheim PA, Nesrallah G, Garg AX, Suri R; Daily Hemodialysis Study Group London Health Sciences Centre. Minutes to recovery after a hemodialysis session: a simple health-related quality of life question that is reliable, valid, and sensitive to change. Clin J Am Soc Nephrol. 2006 Sep;1(5):952-9. doi: 10.2215/CJN.00040106. Epub 2006 Jul 6. PMID 17699312

DOCUMENTS (2):
  • Study Protocol (2018-06-13): https://cdn.clinicaltrials.gov/large-docs/43/NCT03504943/Prot_000.pdf
  • Informed Consent Form (2018-06-13): https://cdn.clinicaltrials.gov/large-docs/43/NCT03504943/ICF_001.pdf